CLINICAL TRIAL: NCT02703064
Title: To Study the Efficacy and Safety of Furocyst in Poly Cystic Ovary Syndrome Patients (PCOS)
Brief Title: Furocyst - Poly Cystic Ovary Syndrome Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chemical Resources (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Protocol No. CR-PCOS/1-15
Record Dates: First submitted 2015-09-29; First posted 2016-03-09 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2016-08

CONDITIONS: PCOS
Keywords: Furocyst; PCOS

STUDY DESIGN:
Intervention Model Description: open level
Oversight: Data Monitoring Committee: No

ARMS (1):
- Furocyst (Experimental): Furocyst 500mg capsule, BD
  Interventions: Dietary Supplement: Furocyst

INTERVENTIONS:
Dietary Supplement: Furocyst — Furocyst caps BD
  Other Names: Standardized fenugreek extract

SUMMARY:
Poly cystic ovary syndrome (PCOS) is the most common endocrine disorder in women of reproductive age, affecting approximately 5%-10% of all females worldwide . PCOS is a hormonal disorder that involves multiple organ systems within the body. Its cardinal features are Hyperandrogenism and polycystic ovary (PCO) morphology. Women with PCOS may complains about irregular menstrual periods or heavy menstrual bleeding, infertility, excessive growth of coarse facial and body hair, obesity, oiliness of the skin, seborrhea, and cystic acne.

DETAILED DESCRIPTION:
The symptoms of PCOS are anovulation, resulting in irregular menstruation (amenorrhea and oligomenorrhea) ovulation-related infertility, and polycystic ovaries, often associated with obesity, Type 2 diabetes, and high cholesterol levels. The level of serum insulin and insulin resistance are higher in women with PCOS (Hyperinsulinemia).Insulin resistance, defined as the decreased insulin mediated glucose utilization it is more common in women with PCOS up to 50 % in both obese and non obese women . It has also been recognized that some women with this syndrome will have PCO without clinical evidence of androgen excess, but will display evidence of ovarian dysfunction .

It is believed to be that, the Hyperinsulinemia of PCOS stimulates the androgens production and increase the activity by decreasing the sex hormone binding globulin (SHBG) thus increasing the free active testosterone level and by the activating the cytochrome P 450 C 17 alpha enzymatic system that controls androgens production.

The diagnosis of PCOS is based on Hyperandrogenism and chronic anovulation in the absence of specific pituitary or adrenal disease , and have disrupted ovulatory function with chronic oligomenorrhea (cycle length > 35 day) or amenorrhea (cycle length > 12 week) and typical appearance of polycystic ovaries by ultrasound according to the criteria of the Rotterdam consensus meeting 2003 for diagnosis of PCOS. The different diagnostic tests needed to adequately assess for the possibility of PCOS e.g. Pregnancy test, TSH level (for Hyperthyroidism), Prolactin test (for Hyperprolactinemia), Total testosterone (for ovarian tumor) and some tests forevaluating the insulin resistance syndrome in women: Waist circumference (>88 cm), Triglycerides (>150 mg/dL), HDL Cholesterol (<50 mg/dL), Blood pressure (>130/85) and Fasting glucose (>110 mg/dL). Fasting glucose- to- insulin ratio and 2 hour oral glucose tolerance test (2h- OGTT 140 - 199 mg/dL) may be better predictor of insulin resistance .

The management of the PCOS is symptoms specific e.g.

1. Oral contraceptives, periodic progesterone withdrawal for the control of irregular menstruation.
2. Oral contraceptives, Metformin and anti-androgens (Spironolactone) for the

   Hirsutism.
3. Clomiphene citrate, Metformin and thiazolidinediones for infertility. A recent study shown that, the combination of Metformin plus Clomiphene citrate should be considered as the First line treatment for infertile women with PCOS .
4. Metformin and lifestyle modification for the insulin resistance and diabetes mellitus.

All these management options are only for "acute" not for "chronic". The long-term management approach for the PCOS is needed which will be based on management of most affecting factor insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women between 18-45 years of age and BMI less than 42
* Diagnosed with PCOS by Rottadom Criteria
* Adequate hepatic, renal, Cardiac and hematological functions.
* Patients willing to Participate and give informed consent in writing as well as in audio-visual form for the study.
* Stable weight for last two months (Change of weight<3kg)

Exclusion Criteria:

* Male
* Post menopausal women
* Women with hysterectomy
* Hyperprolactinemia
* Patients with congenital adrenal hyperplasia
* Patients suffering from Cushing's syndrome
* Acute or chronic Medical illness including Hepatic, Cardiac or renal insufficiency, COPD,Gastrointestinal Disorders
* Uncontrolled Hypertensive or known Diabetics on drugs
* Use of oral contraceptives or HRT for last three months
* Smoking or drug addicts or with psychiatric illness
* Patients diagnosed with androgen secreting tumors.
* Patients with thyroid dysfunction (T3, T4 level is higher than that in normal women of reproductive age)
* Patients with Hypo-gonadotropic and Hypo-gonadism (central origin of ovarian dysfunction)
* Pregnant or lactating mothers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Reduction in Overian volume & Number of overian Cysts | 12 weeks

SECONDARY OUTCOMES:
Restoration of normal menstrual cycle | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pushpalata Sankhwar, M.S., Principal Investigator — Dept of Obs & Gynae,King George's Medical University, Lucknow, UP, India
Locations (1):
- Dept of Obs & Gynae, King George's Medical University, Lucknow, UP, India, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polson DW, Adams J, Wadsworth J, Franks S. Polycystic ovaries--a common finding in normal women. Lancet. 1988 Apr 16;1(8590):870-2. doi: 10.1016/s0140-6736(88)91612-1. PMID 2895373